CLINICAL TRIAL: NCT02475278
Title: Phase II, Single Arm, Open Label Trial for Serologic Assay Validation, Proficiency Testing, Safety and Immunogenicity of the Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine
Brief Title: Serologic Assay Validation, Proficiency Testing, Safety and Immunogenicity of Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NOR-210; U1111-1165-3548 (Registry Identifier: WHO)
Record Dates: First submitted 2015-02-24; First posted 2015-06-18 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Norovirus; Healthy Participants
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NoV Vaccine (Experimental): Norovirus GI.1/GII.4 bivalent Virus-Like Particle (VLP) vaccine (NoV Vaccine) (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP, adjuvanted with 500 µg aluminum hydroxide), intramuscular (IM) injection, once on Day 1.
  Interventions: Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine

INTERVENTIONS:
Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine — Norovirus GI.1/GII.4 bivalent VLP vaccine adjuvanted with aluminum hydroxide for IM injection

SUMMARY:
The purpose of this study is to collect serum samples to evaluate serologic assays and to establish proficiency panels for serologic assays used for assessment of post vaccination immune response after intramuscular (IM) vaccination with Norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called Norovirus GI.1/GII.4 bivalent Virus-Like Particle Vaccine (NoV Vaccine). The purpose of this study is to collect serum samples to evaluate serologic assays and to establish proficiency panels for serologic assays used for assessment of post vaccination immune response after intramuscular (IM) vaccination with the NoV vaccine. The validation and proficiency testing of the immunogenicity assays is required to support the NoV Vaccine development program. This study also looked at side effects in people who were administered a single dose of the NoV vaccine.

The study enrolled 50 patients. All participants received one dose of the NoV vaccine via intramuscular injection.

Participants were asked to record any symptoms that may be related to the vaccine or the injection site in a diary card for 7 days after receiving the vaccination.

This single-centre trial was conducted in the United States. The overall time to participate in this study was 183 days. Participants made 4 visits to the clinic, and were contacted by telephone 183 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 49 years, inclusive.
2. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
3. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Can comply with trial procedures and are available for the duration of follow-up.
5. Body weight of ≥50kg (110lbs).
6. Body mass index (BMI) <35.

Exclusion Criteria:

1. Has a history of acute gastroenteritis (AGE) within 14 days of enrollment.
2. Has previously been exposed to an experimental Norovirus (NoV) Vaccine.
3. Has received any inactivated vaccines within 14 days or any live vaccines for 28 days prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine administration.
4. Has contraindications, warnings and/or precautions to vaccination with the NoV Vaccine as specified within the investigator brochure.
5. Has known hypersensitivity or allergy to any of the NoV Vaccine components (including excipients).
6. Has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.
7. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g. Guillain-Barré syndrome).
8. Has history or any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
9. Has known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1.
   3. Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the investigational vaccine or planned administration during the trial (consider whether applicable as an exclusion criterion or criterion for delay).
   4. Receipt of immunostimulants within 60 days prior to Day 1.
   5. Receipt of parenteral, epidural or intra-articular immunoglobulin preparation, blood products, and/or plasma derivates within 3 months prior to Day 1 or planned during the full length of the trial.
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Genetic immunodeficiency.
10. Has abnormalities of splenic or thymic function.
11. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
12. Has any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
13. Is participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
14. Is involved in the trial conduct or their first degree relatives.
15. Has history of substance or alcohol abuse within the past 2 years.
16. Females who are pregnant or breastfeeding.
17. If female of childbearing potential, sexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry:

    1. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
    2. Acceptable birth control methods are defined as one or more of the following:

    i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).

    ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.

    iii. Intrauterine device (IUD). iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
18. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" through to 6 months after receipt of investigational vaccine. In addition, they must be advised not to donate ova during this period.
19. Any positive or indeterminate pregnancy test.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Benchmark Research Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Atmar RL, Ettayebi K, Neill FH, Braun RP, Sherwood J, Ramani S, Estes MK. Correlation of Genogroup I, Genotype 1 (GI.1) Norovirus Neutralizing Antibody Levels With GI.1 Histo-Blood Group Antigen-Blocking Antibody Levels. J Infect Dis. 2024 Dec 16;230(6):1376-1379. doi: 10.1093/infdis/jiae311. PMID 38864524
- [Derived] Atmar RL, Ettayebi K, Ayyar BV, Neill FH, Braun RP, Ramani S, Estes MK. Comparison of Microneutralization and Histo-Blood Group Antigen-Blocking Assays for Functional Norovirus Antibody Detection. J Infect Dis. 2020 Feb 18;221(5):739-743. doi: 10.1093/infdis/jiz526. PMID 31613328
- [Derived] Atmar RL, Cramer JP, Baehner F, Han C, Borkowski A, Mendelman PM. An Exploratory Study of the Salivary Immunoglobulin A Responses to 1 Dose of a Norovirus Virus-Like Particle Candidate Vaccine in Healthy Adults. J Infect Dis. 2019 Jan 9;219(3):410-414. doi: 10.1093/infdis/jiy529. PMID 30203081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 26 February 2015 to 9 September 2015.
Pre-assignment Details: Healthy volunteers were enrolled in 1 treatment group and received a single dose of NoV Vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP, adjuvanted with 500 µg aluminum hydroxide).
Period: Overall Study
Arm/Group | NoV Vaccine
Started | 50
Completed | 48
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black Or African American | 14
  White | 36
Region of Enrollment [Number; unit: participants]
  United States | 50
Height [Mean (Standard Deviation); unit: cm] | 171.42 (9.115)
Weight [Mean (Standard Deviation); unit: kg] | 79.08 (13.864)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.88 (4.025)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Samples Obtained on Day 8 for Assessment of Seropositivity for Both Anti-NoV GI.1 VLP and GII.4 VLP Antibodies
Description: Serum samples were obtained for assay validation of the pan-Ig enzyme-linked immuno-sorbent assay (ELISA) and the histoblood group antigen (HBGA) binding assay. The number of participants with assessments for both the GI.1 VLP and GII.4 VLP antibodies and by both the pan-Ig ELISA and the HBGA binding assay, and with values available at Baseline and Day 8 are reported.
Time Frame: Day 8
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
participants | 48

2. Primary Outcome: Number of Participants With Serum Samples Obtained on Day 15 for Assessment of Seropositivity for Both Anti-NoV GI.1 VLP and GII.4 VLP Antibodies
Description: Serum samples were obtained to establish proficiency panels for the pan-Ig ELISA and the HBGA binding assay. The number of participants with assessments for both the GI.1 VLP and GII.4 VLP antibodies and by both the pan-Ig ELISA and the HBGA binding assay, and with values available at Baseline and Day 15 are reported.
Time Frame: Day 15
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
participants | 48

3. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) by Maximum Severity
Description: Safety assessment included collection of solicited local AEs for 7 days following vaccination (including the day of vaccination) by using diary cards. Solicited local injection site AEs are defined as pain, erythema (redness), induration and swelling. Pain is summarized as either none or any, where 'any' will be broken down into the following severity categories: mild, moderate, severe. Erythema, swelling and induration are recorded as yes or no, where the definition of 'yes' is any area ≥2.5 cm; and 'yes' is further broken down into the following severity categories: ≥2.5 cm - ≤5.0 cm (mild intensity), >5.0 cm - ≤ 10.0 cm (moderate intensity), >10.0 cm severe intensity). Injection site AEs are presented as the percentage of participants experiencing a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: Days 1 through 7
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
percentage of participants
  Pain, Any | 54.0
  Pain, Mild | 44.0
  Pain, Moderate | 10.0

4. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Maximum Severity
Description: Safety assessment included collection of solicited systemic AEs for 7 days following vaccination (including the day of vaccination) by using diary cards. Solicited systemic AEs are defined as headache, fatigue, myalgia, arthralgia, vomiting and diarrhea and are summarized as either none or any, where 'any' will be broken down into the following severity categories: mild, moderate, severe. Solicited systemic AEs are presented as the percentage of participants experiencing a solicited systemic AE, by AE, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: Days 1 through 7
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
percentage of participants
  Headache, Any | 24.0
  Headache, Mild | 18.0
  Headache, Moderate | 6.0
  Fatigue, Any | 34.0
  Fatigue, Mild | 30.0
  Fatigue, Moderate | 4.0
  Myalgia, Any | 12.0
  Myalgia, Mild | 12.0
  Arthralgia, Any | 6.0
  Arthralgia, Mild | 6.0
  Vomiting, Any | 2.0
  Vomiting, Mild | 2.0
  Diarrhea, Any | 12.0
  Diarrhea, Mild | 10.0
  Diarrhea, Moderate | 2.0

5. Secondary Outcome: Percentage of Participants With Elevated Daily Oral Temperature
Description: Safety assessment included measurement of body temperature for 7 days following vaccination (including the day of vaccination) by using diary cards. Participants recorded the highest body temperature observed each day in a daily diary. The highest body temperature measurement per participant across Day 1 to Day 7 was categorized as fever present (≥100.4ºF, ≥38ºC) or fever absent (<100.4ºF, <38ºC).
Time Frame: Days 1 to 7 days after vaccination
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
percentage of participants | 0.0

6. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs) by Maximum Severity
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study. Unsolicited AEs are presented as the percentage of participants experiencing at least one AE, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: Days 1 through 28
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
percentage of participants
  Unsolicited Adverse Events, Any | 22.0
  Unsolicited Adverse Events, Mild | 14.0
  Unsolicited Adverse Events, Moderate | 6.0
  Unsolicited Adverse Events, Severe | 2.0

7. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events
Description: A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Day 1 up to Day 183
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
percentage of participants | 2.0

8. Primary Outcome: Number of Participants With Serum Samples Obtained on Day 29 for Assessment of Seropositivity for Both Anti-NoV GI.1 VLP and GII.4 VLP Antibodies
Description: Serum samples were obtained to establish proficiency panels for the pan-Ig ELISA and the HBGA binding assay. The number of participants with assessments for both the GI.1 VLP and GII.4 VLP antibodies and by both the pan-Ig ELISA and the HBGA binding assay, and with values available at Baseline and Day 29 are reported.
Time Frame: Day 29
Population: Safety Analysis Set, all participants who received the trial vaccine (NoV Vaccine).
Measure: Number; unit: participants
Arm/Group | NoV Vaccine
Number analyzed (Participants) | 50
participants | 46

ADVERSE EVENTS:
Time Frame: Unsolicited AEs 28 days after vaccination (Day 1 to 28) and Serious Adverse Events (SAEs) throughout the trial (Up to Day 183).
Description: At each visit the investigator documented any occurrence of AEs. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. Non-serious unsolicited AEs reported below. Non-serious solicited AEs reported in the outcome measure section.
Arm/Group | NoV Vaccine
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NoV Vaccine (N=50)
Unevaluable event (General disorders) | 1 — One participant was reported as having "unknown event leading to hospitalization".
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NoV Vaccine (N=50)
Rhinitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.